CLINICAL TRIAL: NCT06981507
Title: Evaluation of the Effect of MARPE on Speech
Acronym: MARPE-Speech
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Necmettin Erbakan Üniversitesi (Other)
Responsible Party: Principal Investigator, KAZIM KAAN YILDIZ, Research Assistant, Konya Necmettin Erbakan Üniversitesi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2025536
Record Dates: First submitted 2025-05-01; First posted 2025-05-20 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Evaluation of Speech Characteristics Following MARPE Treatment in Patients With Maxillary Transverse Deficiency
Keywords: MARPE, Palatal Expansion, Orthodontics, Speech, Acoustic Analysis, Maxillary Transverse Deficiency
MeSH Terms: conditions — Speech

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MARPE Intervention Group (Experimental)
  Interventions: Device: MARPE (Miniscrew-Assisted Rapid Palatal Expansion)

INTERVENTIONS:
Device: MARPE (Miniscrew-Assisted Rapid Palatal Expansion) — MARPE (Miniscrew-Assisted Rapid Palatal Expansion) is an orthodontic expansion technique that uses a palatal expander anchored with miniscrews inserted into the palatal bone. The device applies lateral force to widen the maxilla skeletally in patients with transverse maxillary deficiency. In this study, all participants will receive MARPE treatment as part of their orthodontic management, and its potential effects on speech will be evaluated over time.

SUMMARY:
This study investigates the effects of Miniscrew-Assisted Rapid Palatal Expansion (MARPE) on speech characteristics in adolescent and young adult patients.

While MARPE is a widely used orthodontic procedure for treating maxillary transverse deficiency, its potential impact on speech production has not been thoroughly evaluated. The aim of this study is to assess whether MARPE treatment causes any temporary or long-term changes in speech patterns using acoustic and perceptual analysis methods.

DETAILED DESCRIPTION:
This prospective clinical study aims to evaluate how Miniscrew-Assisted Rapid Palatal Expansion (MARPE) affects speech in adolescents and young adults with skeletal maxillary transverse deficiency.

Speech production relies on precise palatal anatomy and oral resonance. Since MARPE modifies the palatal structure through skeletal expansion, it may influence articulation and acoustic properties of speech. Despite its increasing use in orthodontics, the potential speech-related side effects of MARPE remain largely unexplored.

Participants aged 13-25 will undergo MARPE treatment as part of their standard orthodontic care. Speech recordings will be taken at three time points: before expansion (baseline), immediately after the active expansion phase, and after the retention period. Acoustic analysis and standardized perceptual speech evaluations will be conducted to detect any phonetic, articulatory, or resonance-related changes.

The results will help clinicians better understand the functional implications of MARPE on speech and provide guidance for counseling patients before treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Class I malocclusion
* Presence of maxillary transverse deficiency
* Young adult patients aged 15 to 18 years
* No history of systemic disease, cleft lip/palate, or speech disorders
* No history of previous orthodontic treatment

Exclusion Criteria:

* Patients with any systemic disease
* Patients who smoke
* Patients with poor oral hygiene
* Patients with cooperation difficulties
* Patients with mental retardation or cognitive impairment

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Speech Changes After MARPE Treatment | Baseline and 1 month after expansion

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Faculty of Dentistry, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including speech evaluation results and relevant demographic variables, will be shared with qualified researchers upon reasonable request. Data will be made available starting 6 months after publication of study results and will remain accessible for 3 years. Requests must be submitted via institutional email and will require a data use agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Data and supporting documents (Study Protocol and Statistical Analysis Plan) will be available beginning 6 months after the publication of study results and will remain accessible for 3 years.
Access Criteria: Access to de-identified individual participant data and supporting documents will be granted to qualified researchers upon reasonable request. Requestors must provide a methodologically sound proposal and sign a data use agreement. Data will be shared via secure institutional channels following approval by the principal investigator.

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27463698/